CLINICAL TRIAL: NCT06933316
Title: The Effect of Family-Integrated Care Model on Infant and Toddler Health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoqi Lin (Other)
Responsible Party: Sponsor-Investigator, Xiaoqi Lin, Chief Physician, Nanchong Maternal and Child Health and Family Planning Service Center
Organization: Nanchong Maternal and Child Health and Family Planning Service Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No. 2024058
Record Dates: First submitted 2025-04-09; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Family Caregiving; Infant Health; Growth; Nutrition; Cognition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Other): the intervention group received additional FIC-based care, including individualized health plans, education, daily care guidance, dietary recommendations, micronutrient supplementation, early intervention, growth monitoring, and vaccination support.
  Interventions: Other: the intervention group
- the control group (Other): The control group received routine health guidance
  Interventions: Other: the control group

INTERVENTIONS:
Other: the intervention group — the intervention group received additional FIC-based care, including individualized health plans, education, daily care guidance, dietary recommendations, micronutrient supplementation, early intervention, growth monitoring, and vaccination support.
  Arms: the intervention group
Other: the control group — Infants receive routine healthcare guidance provided by pediatric healthcare professionals. This includes regular check-ups scheduled via phone appointments, general health consultations, vaccinations according to regulations, and tailored feeding and parenting guidance based on examination results.
  Arms: the control group

SUMMARY:
The FIC model effectively promotes infant growth, improves nutrition, reduces disease risk, and supports early cognitive and psychological development while enhancing parental caregiving skills, demonstrating strong clinical value.

DETAILED DESCRIPTION:
This study explored the effects of the family-integrated care (FIC) model on growth, nutrition, disease incidence, and early cognitive and psychological development in infants aged 6-18 months. A total of 158 full-term infants were randomly assigned to an intervention group (n=79) or a control group (n=79). The control group received routine health guidance, while the intervention group received additional FIC-based care, including individualized health plans, education, daily care guidance, dietary recommendations, micronutrient supplementation, early intervention, growth monitoring, and vaccination support. Outcomes assessed at baseline and six months post-intervention included growth indices (weight, height, head circumference), nutritional markers (hemoglobin, vitamin D), disease incidence (respiratory infections, gastrointestinal dysfunction, eczema), and Bayley Scales of Infant Development scores. Parental adherence, satisfaction, and caregiving competency were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born in our hospital who undergo regular check-ups in the pediatric healthcare department.
2. Age between 6 and 18 months.
3. Complete and comprehensive clinical data.
4. Full-term birth.
5. Families voluntarily participate and sign informed consent.
6. Parents are in good health and have time to accompany their children daily.

Exclusion Criteria:

1. Congenital diseases.
2. Infectious diseases.
3. Familial hereditary diseases.
4. Abnormal conditions during pregnancy or perinatal period.
5. Missing clinical data.
6. No willingness to participate in this study.
7. Abnormal physical or intellectual development of the infant.
8. Intellectual disabilities of the guardians. -

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2022-03-13 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
The Effect of Family-Integrated Care Model on Infant and Toddler Health Promotion | 5 months
  The FIC model effectively promotes infant growth, improves nutrition, reduces disease risk, and supports early cognitive and psychological development while enhancing parental caregiving skills, demonstrating strong clinical value.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Maternal and Child Health and Family Planning Service Center, Nanchong, China